CLINICAL TRIAL: NCT04694378
Title: Relationship Between Right Ventricular Free Wall Longitudinal Strain and Stroke Volume Index by Thermodilution in Patients Undergoing Cardiac Surgery
Brief Title: Relationship Between Strain and Stroke Volume in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2020-12-16; First posted 2021-01-05 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Right Ventricular Dysfunction; Stroke Volume Index; Longitudinal Heart Strain
Keywords: Echocardiography; Coronary artery bypass graft; Thermodilution
MeSH Terms: conditions — Ventricular Dysfunction, Right

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients undergoing coronary artery bypass grafting up tp 30% will develop postoperative right ventricle dysfunction. Its imperative for the physician to fully understand the severity of this complication in order to perform an early diagnosis and carry out the appropriate treatment.

Aim:

Investigate the correlation between echocardiographic measurements and hemodynamic changes at different time points in patients undergoing coronary artery bypass graft surgery

Hypothesis:

1. Weak correlation between echocardiographic measurements and hemodynamic changes during coronary artery bypass graft surgery
2. Echocardiographic measurements would change across different time points during surgery independent of hemodynamic values.

ELIGIBILITY:
Inclusion Criteria:

- Elective coronary artery bypass graft patients who require pulmonary catheter placement for intraoperative monitoring.

Exclusion Criteria:

* Patients with contraindication to Swan-Ganz catheter placement,
* Pre-existing atrial arrhythmias,
* Patients with moderate and/or severe mitral/tricuspid valve stenosis or regurgitation
* Patients with contraindication to transesophageal echocardiogram probe placement (i.e. esophageal stenosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients older that 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Change of right ventricular function during CABG assessed by right heart strain (%) | during CABG surgery
  Assessing the change of RV function during CABG surgery using right heart strain as a percentage of change between RV shortening and RV end diastolic length.
Change of right ventricular function during CABG assessed by stroke volume index (mL/m2) | during CABG surgery
  Assessing the change of RV function during CABG surgery using stroke volume index. Stroke volume index measurement as millilitres per square meter (ml/m2)

SECONDARY OUTCOMES:
Change in cardiac output measured with Swan-Ganz during CABG | during CABG surgery
  Cardiac output (L/min) measured with the thermodilution technique

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No